CLINICAL TRIAL: NCT02961283
Title: A Phase 1, Open-label, Dose-finding and Cohort Expansion Study of ASN003 in Subjects With Advanced Solid Tumors
Brief Title: Study of ASN003 in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: reformulation
Sponsor: Asana BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASN003-101
Record Dates: First submitted 2016-10-25; First posted 2016-11-10 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Neoplasms; Melanoma; Colorectal Neoplasm; Carcinoma, Non-small Cell Lung
Keywords: BRAF Kinases; PIK3CA protein, human
MeSH Terms: conditions — Neoplasms; Melanoma; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- ASN003 Dose Escalation (Experimental): Multiple ascending doses of ASN003 will be administered to determine the maximum tolerated dose (MTD).
  Interventions: Drug: ASN003 ascending doses
- ASN003 MTD - BRAFv600 melanoma (Experimental): ASN003 administered at the MTD in subjects with BRAF v600 mutated metastatic melanoma
  Interventions: Drug: ASN003 MTD
- ASN003 MTD - BRAFv600 colon or lung cancer (Experimental): ASN003 administered at the MTD in subjects with BRAFv600 mutated metastatic colorectal or non-small cell lung cancer.
  Interventions: Drug: ASN003 MTD
- ASN003 MTD - PIK3 pathway mutated cancers (Experimental): ASN003 administered at the MTD in subjects who have mutations in PI3 kinase or loss of PTEN.
  Interventions: Drug: ASN003 MTD

INTERVENTIONS:
Drug: ASN003 ascending doses
  Arms: ASN003 Dose Escalation
Drug: ASN003 MTD — The highest safe and well tolerated dose selected from the doses tested in Part A of the study.
  Arms: ASN003 MTD - BRAFv600 colon or lung cancer; ASN003 MTD - BRAFv600 melanoma; ASN003 MTD - PIK3 pathway mutated cancers

SUMMARY:
The study is divided into two parts. The first part of the study will test various doses of ASN003 to find out the highest safe dose to test in three specific groups.

The second part of the study will test how well ASN003 can control cancer. Subjects will be enrolled into one of three groups.

Group 1: metastatic or recurrent melanoma with documented BRAFV600 mutation (n=20 evaluable patients) Group 2: metastatic colorectal cancer (CRC), or advanced non-small cell lung cancer (NSCLC) with documented BRAFV600 mutation (n=14 evaluable patients) Group 3: advanced solid tumors with documented PI3K pathway alterations (PIK3CA mutation or PTEN loss) (n=14 evaluable patients)

DETAILED DESCRIPTION:
The study will be conducted in two parts. Part A is a dose escalation study to determine a safe and tolerable dose of ASN003 for subjects with advanced solid tumors. Part A will also characterize the pharmacokinetics and pharmacodynamics of ASN003 through blood sampling and optional biopsies.. Part B will only enroll subjects in three groups:

Group 1: subjects who have metastatic or recurrent melanoma with the BRAFv600 mutation.

Group 2: subjects who have advanced or metastatic non-small cell lung cancer, or colorectal cancer with the BRAFv600 mutation.

Group 3: subjects who have advanced or metastatic cancers with phosphatidylinositide 3-kinases (PI3K) mutations, or phosphatase and tensin homolog (PTEN) loss mutation. Subjects will be treated with the highest safe and tolerable dose determined in Part A of the study to determine preliminary efficacy. Subjects may continue to receive ASN003 for up to 1 year in the absence of severe side effects or disease progression.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent obtained prior to any study-related procedures.
* Eastern Cooperative Oncology Group Performance Status: 0-1
* Part A only: Histologically or cytologically confirmed metastatic and/or advanced solid tumors with documented progressive disease for whom no further standard therapy is indicated.
* Part B only: 5. Histologically or cytologically confirmed, molecularly selected (i.e. BRAFV600 positive and/or PI3K mutation positive) advanced solid tumors. Prior molecular characterization should be based using a regulatory approved assay or analytically validated assay.

  * Group 1: BRAFV600 positive metastatic or recurrent melanoma after failure of prior treatment with standard therapy such as a checkpoint inhibitor and an approved B-RAF inhibitor (vemurafenib or dabrafenib)
  * Group 2: BRAFV600 positive metastatic colorectal carcinoma (CRC), or advanced non-small cell lung carcinoma (NSCLC) after failure of at least two lines of prior standard therapy or for whom no further standard therapy is indicated.
  * Group 3: Advanced solid tumors with PI3K pathway alterations (PIK3CA mutation or PTEN loss) after failure of at least one line of prior standard therapy or for whom no further standard therapy is indicated. Prior treatment may not include inhibitors of the PI3K pathway.
* Screening hematology values of the following: absolute neutrophil count ≥ 1000/μL, platelets ≥ 100,000/μL, hemoglobin ≥ 10 g/dL (without transfusion support);
* Screening chemistry values of the following: alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 3.0 × upper limit of the normal reference range (ULN), total bilirubin ≤ 2 × ULN, creatinine ≤ 1.5 × ULN, fasting blood glucose < 140 mg/dL, hemoglobin A1C ≤ ULN, albumin ≥ 2.8 g/dL.
* Screening fasting lipid panel: LDL cholesterol < 190 mg/dL, triglycerides < 300 mg/dL
* Subject is willing and able to comply with all protocol required visits and assessments, including biopsy if assigned to the MTD expansion cohort;

Exclusion Criteria:

* Have received prior chemotherapy, other investigational therapy, or major surgery within 4 weeks of Day 1;
* Have received oral anti-cancer therapy with oral tyrosine kinase inhibitors within 14 days or 5 half-lives, whichever is longer.
* Have received prior treatment with monoclonal antibodies within 6 weeks of first dose of Day 1;
* Subject has received a live virus vaccine within the previous 8 weeks.
* Have known central nervous system metastasis or primary tumor (Part A). Previously-treated, CNS metastasis is permitted in Part B. CNS metastasis must be small, discrete metastasis; stable for at least 30 days without the need for concomitant prednisone for symptom management. No leptomeningeal disease is allowed. Is receiving therapeutic doses of corticosteroids (>20 mg prednisone daily or equivalent);
* Has a serious concurrent medical condition such as:

  * history of Diabetes Mellitus, type 1 or type 2,
  * known autoimmune disease, known bleeding diathesis, history of congestive heart failure New York Heart Association (NYHA) class III or IV;
  * uncontrolled hypertension (systolic BP ≥ 139 mmHg or diastolic BP ≥ 89 mmHg) at screening, despite optimal antihypertensive therapy,
  * clinically significant heart disease including but not limited to: myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or known cardiac ejection fraction measurement of < 50 %;
  * history or family history of long QT syndrome; 12-Lead electrocardiogram (ECG) abnormalities considered by the investigator to be clinically significant or QTcF ≥ 450 milliseconds, regardless of clinical significance, at screening. Abnormal ECG may be confirmed with one repeat assessment. For subjects with QTcF ≥ 450 msec on initial ECG, the mean of the two QTcF assessments will determine eligibility;
  * uncontrolled psychiatric illness;
  * serious persistent infection within 14 days prior to the start of study medication;
  * known gastrointestinal disease or condition which may affect the absorption of ASN003;
  * known active or symptomatic viral hepatitis, chronic liver disease or liver cirrhosis;
  * known glaucoma or other pre-existing ocular conditions that may put the patient at risk for ocular toxicities.
  * any known condition or situation which may put the patient at significant risk, may confound the study results, or may interfere significantly with subject's participation in the study
* Female subjects who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-10; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Part A: Determine the maximum tolerated dose (MTD) of ASN003 | First 21 days
  The MTD will be determined by evaluating the number of subjects with treatment related dose limiting toxicity. This is the primary endpoint of Part A
Part B: evaluates the preliminary efficacy of ASN003 in subjects with selected BRAF and PI3 kinase mutated cancers | Up to 1 year
  Evaluation of the overall disease status using the RECIST 1.1 terms of complete response, partial response, stable disease, and progressive disease. This is the primary endpoint for Part B

SECONDARY OUTCOMES:
Calculate the Pharmacokinetic Area Under the Curve | First 22 days
  A plot of the concentration of ASN003 in blood plasma over time.
Calculate the Pharmacokinetic Maximum Concentration | First 22 days
  The peak plasma concentration of ASN003
Calculate the Pharmacokinetic Half-life | First 22 days
  The time required for ASN003 to lose half of its pharmacologic activity.
Change from baseline in pharmacodynamic biomarkers | Up to 1 year
  Pre-dose and post-dose pharmacodynamic biomarkers in plasma and tumor biopsy will be compared to assess signs of pharmacodynamic activity
Change in the size of measurable tumor lesions | Up to 1 year
  Change from baseline in the sum of the longest dimension in centimeters of each measurable lesion, the presence/absence of lesions that cannot be measured in centimeters, or the presence of new lesions.
Change in the status of non-measurable tumor lesions | Up to 1 year
  Number of subjects that have resolution of non-measurable tumor lesions.
Appearance of new tumor lesions | Up to 1 year
  Number of subjects with new lesions

OTHER OUTCOMES:
Change in tumor mutational status | Up to 1 year
  Tumor biopsy samples will be tested to look for changes

CONTACTS AND LOCATIONS:
Overall Officials: Asana BioSciences, Study Director — Asana BioSciences, LLC
Locations (5):
- United States (5):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - START MidWest, Grand Rapids, Michigan
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No